CLINICAL TRIAL: NCT03160456
Title: Randomised Controlled Trial of Domiciliary Transcutaneous Electrical Stimulation in Obstructive Sleep Apnoea
Brief Title: Domiciliary Transcutaneous Electrical Stimulation in Obstructive Sleep Apnoea
Acronym: TESLA-home
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Collaborators: King's College London (Other); Royal Brompton & Harefield NHS Foundation Trust (Other); King's College Hospital NHS Trust (Other)
Responsible Party: Principal Investigator, Joerg Steier, Consultant Physician, Guy's and St Thomas' NHS Foundation Trust
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Version 1.3 / 22-11-2020; 217448 (Other: IRAS); 18/LO/0638 (Other: REC reference)
Record Dates: First submitted 2017-05-16; First posted 2017-05-19 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Obstructive Sleep Apnea
Keywords: upper airway; genioglossus; CPAP; electrical stimulation; sleep; sleep disordered breathing
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Apnea Syndromes | interventions — Transcutaneous Electric Nerve Stimulation; Continuous Positive Airway Pressure

STUDY DESIGN:
Intervention Model Description: Randomised parallel group controlled clinical trial
Who Masked: Outcomes Assessor
Masking Description: No masking
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transcutaneous electrical stimulation (Experimental): The group of participants receiving continuous transcutaneous electrical stimulation will be trained on the device and settings will be recorded. The device is kept on all night and in the morning taken off with the hydrogel and disconnected. Bi-weekly phone calls and follow up visits at 6- and 12-weeks will be organized. At each visit comfort, compliance and adverse reactions will be recorded. At 12-weeks, the patients will be invited for a repeat assessment including polysomnography/home-based respiratory polygraphy during a night of electrical stimulation. Usage time of the device will be discussed with the patients and recorded.
  Interventions: Device: Transcutaneous electrical stimulation
- Continuous positive airway pressure (usual care) (Active Comparator): Participants who will be randomized to the usual care group will be given their own CPAP device, as previously prescribed. Bi-weekly phone calls and follow up visits at 6- and 12-weeks will be organized. At the last visit, the patients will be studied during a repeat inpatient polysomnography/home-based respiratory polygraphy and the initial assessment will be repeated.
  Interventions: Device: Continuous positive airway pressure

INTERVENTIONS:
Device: Transcutaneous electrical stimulation — The device needs to be started by pressing the 'on' button. Once the device is turned on the current intensity can be increased by pushing the '+' button and lowered by pushing the '-' button. When a comfortable skin sensation is felt the patients should press the '-' button once more. At that time the device stimulates with a low current which is not felt but provides a neuromuscular tone to the muscles whilst asleep. The device is kept on all night and in the morning taken off with the hydrogel and disconnected. Once disconnected it should be turned off by pressing the 'off' button.
  Other Names: TESLA home
  Arms: Transcutaneous electrical stimulation
Device: Continuous positive airway pressure — CPAP will be applied according to usual clinical care, the follow up will be organised in the same way as the active intervention group.
  Other Names: CPAP (usual care)
  Arms: Continuous positive airway pressure (usual care)

SUMMARY:
The aim of this study is to assess the efficacy of transcutaneous electrical stimulation of the pharyngeal dilator muscles in patients with obstructive sleep apnoea in the community compared to usual care, and follow the patients for three months, as well as to assess compliance of non-invasive electrical stimulation of the upper airway dilator muscles in obstructive sleep apnoea patients over time and evaluate the control of symptoms and improvement in quality of life.

DETAILED DESCRIPTION:
Obstructive sleep apnoea is highly prevalent, with the obesity epidemic increasing the problem. The best treatment for uncomplicated and moderate-severe OSA remains CPAP therapy. However, long-term adherence to treatment with CPAP is poor and there are few alternatives. Electrical stimulation of the dilator muscles of the upper airway has been shown to reduce nocturnal apnoeas significantly using an invasive approach, hypoglossal nerve stimulation, as well as by non-invasive transcutaneous stimulation. Although non-invasive transcutaneous stimulation may not be as effective as CPAP therapy in many OSA patients it could be an important option to treat some of the large number of patients who fail CPAP and might also be of use in those whose OSA is not judged sufficiently severe to warrant CPAP.

The investigators propose a study to use a transcutaneous electrical stimulation device in selected patients with OSA who do not tolerate CPAP therapy following assessment of the upper airway. Participants will undergo a baseline sleep study (polysomnography/home-based respiratory polygraphy). Following minimisation for gender (male/female) and OSA severity (mild/moderate-severe) they will be randomised into active treatment arm (transcutaneous electrical stimulation) or usual care (ongoing CPAP therapy). Patients will be treated over a period of 3-months in the community, re-assessed (including polysomnography/home-based respiratory polygraphy) and the results will be compared against usual care, ongoing CPAP therapy. This study will help to prepare a definitive multi-centre randomized controlled trial using the non-invasive method of upper airway stimulation in OSA.

The primary aim of this study is to assess efficacy and generate an accurate sample size estimation, test the subjective willingness of patients to use and objectively determined compliance with the treatment over a long period, as well as to specify the drop-out rate. The improvement in sleep apnoea will be the primary outcome measures. The symptomatic response, feasibility of the method, including compliance, comfort, adverse events, will be the secondary outcome measure. An ad-hoc analysis will be performed in the responder group (improvement in the apnoea-hypopnea index (AHI) by >50% from baseline OR improvement in the 4% oxygen-desaturation index (ODI) >25% from baseline OR AHI/4%ODI <5/hour at follow up).

ELIGIBILITY:
Inclusion Criteria:

* mild-moderate OSA (AHI 5-35/hour)
* difficulties with or failed CPAP and/or withdrawn from standard care (CPAP <4hours/night)
* Body mass index (BMI) 18.5-32 kg/m2
* No significant anatomical obstruction in the upper airway (e.g. normal sized tonsils).

Exclusion Criteria:

* No OSA (AHI <5/h)
* Severe obstructive sleep apnoea (AHI>35/hour)
* Exclusively postural sleep apnoea
* isolated Rapid-Eye-Movement (REM) sleep associated OSA
* Cachexia (BMI <18.5 kg/m2)
* Obesity (BMI >32 kg/m2)
* Hypercapnic respiratory failure (pCO2>6.5 kPa)
* Features of obesity hypoventilation syndrome (elevated bicarbonate, HCO3- >28mmol/L).
* enlarged tonsils (size 3-4)
* polyps and adenoids
* neuromuscular disease
* hypoglossal nerve palsy
* abnormal pulmonary function tests
* severe pulmonary hypertension
* valvular heart disease
* heart failure (New York Heart Association, NYHA III-IV)
* myocardial infarction and significant cardiac arrhythmias
* uncontrolled hypertension
* active psychiatric disease
* co-existing non-respiratory sleep disorder
* significant metal implants or cardiac/other pacemakers.
* facial hair that affects the correct placement of the hydrogel patch
* endoscopically identified contraindication to upper airway stimulation (multi-level obstruction)

These criteria are consistent with our experience from previous trials using transcutaneous electrical stimulation in OSA and likely to identify potential responders; these criteria are also similar to those from trials using hypoglossal nerve stimulation.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2018-06-18 (Actual); Primary Completion 2023-02-08 (Actual); Study Completion 2023-05-05 (Actual)

PRIMARY OUTCOMES:
Apnoea Hypopnoea Index | 3 months
  AHI

SECONDARY OUTCOMES:
Epworth Sleepiness Scale | 3 months
  ESS (0-24 points)
Oxygen Desaturation Index | 3 months
  4%ODI (x hour-1)
Usage of treatment | 3 months
  Usage per night (average hours)
Compliance with treatment | 3 months
  Percentage of nights used (%)
Acceptance of device | 3 months
  Visual analogue scale (points, 0-10)
Sleep related quality of life | 3 months
  FOSQ
Snoring | 3 months
  Percentage of the night (%)
Genioglossus contraction | 3 months
  Ultrasound (thickness, mm)
General quality of life | 3 months
  EQ-5D
Anatomy of upper airway | at baseline
  Endoscopically identified diameter (mm)

OTHER OUTCOMES:
Responder rate | 3 months
  Reduction in AHI by more than 50% and / or to below 5/hour

CONTACTS AND LOCATIONS:
Overall Officials: Joerg Steier, MD, PhD, Principal Investigator — Guy's and St Thomas' NHS Foundation Trust; John Moxham, MD, Study Chair — King's College London; Michael I Polkey, PhD, Principal Investigator — Royal Brompton & Harefield NHS Foundation Trust; Kai Lee, MD, Principal Investigator — King's College London NHS Foundation Trust
Locations (1):
- Guy's & St Thomas' NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Yes, upon request to the authors.
Supporting Information: Study Protocol, SAP
Time Frame: The study protocol has been published (Journal of Thoracic Disease 05/2019)
Access Criteria: Upon request
URL: http://jtd.amegroups.com/article/view/29094

REFERENCES:
- [Background] Pengo MF, Steier J. Emerging technology: electrical stimulation in obstructive sleep apnoea. J Thorac Dis. 2015 Aug;7(8):1286-97. doi: 10.3978/j.issn.2072-1439.2014.04.04. PMID 26380757
- [Background] Bisogni V, Pengo MF, De Vito A, Maiolino G, Rossi GP, Moxham J, Steier J. Electrical stimulation for the treatment of obstructive sleep apnoea: a review of the evidence. Expert Rev Respir Med. 2017 Sep;11(9):711-720. doi: 10.1080/17476348.2017.1358619. Epub 2017 Jul 27. PMID 28730908
- [Result] Pengo MF, Xiao S, Ratneswaran C, Reed K, Shah N, Chen T, Douiri A, Hart N, Luo Y, Rafferty GF, Rossi GP, Williams A, Polkey MI, Moxham J, Steier J. Randomised sham-controlled trial of transcutaneous electrical stimulation in obstructive sleep apnoea. Thorax. 2016 Oct;71(10):923-31. doi: 10.1136/thoraxjnl-2016-208691. Epub 2016 Jul 19. PMID 27435610
- [Result] Campbell T, Pengo MF, Steier J. Patients' preference of established and emerging treatment options for obstructive sleep apnoea. J Thorac Dis. 2015 May;7(5):938-42. doi: 10.3978/j.issn.2072-1439.2015.04.53. PMID 26101652
- [Result] Steier J, Seymour J, Rafferty GF, Jolley CJ, Solomon E, Luo Y, Man WD, Polkey MI, Moxham J. Continuous transcutaneous submental electrical stimulation in obstructive sleep apnea: a feasibility study. Chest. 2011 Oct;140(4):998-1007. doi: 10.1378/chest.10-2614. Epub 2011 Mar 31. PMID 21454399
- [Derived] Ratneswaran D, Cheng M, Nasser E, Madula R, Pengo M, Hope K, Schwarz EI, Luo Y, Kaltsakas G, Polkey MI, Moxham J, Steier J. Domiciliary transcutaneous electrical stimulation in patients with obstructive sleep apnoea and limited adherence to continuous positive airway pressure therapy: a single-centre, open-label, randomised, controlled phase III trial. EClinicalMedicine. 2023 Aug 3;62:102112. doi: 10.1016/j.eclinm.2023.102112. eCollection 2023 Aug. PMID 37654667
- See also: Open access link to the first randomised sham-controlled study of TESLA — http://thorax.bmj.com/content/71/10/923.long
- See also: Open access link to a review about invasive and non-invasive electrical stimulation in sleep apnoea — http://jtd.amegroups.com/article/view/2429/5199
- Available data/document: NICE guidance "Hypoglossal Nerve Stimulation": IPG598 — https://www.nice.org.uk/guidance/ipg598 — National Institute for Health and Care Excellence

DOCUMENTS (1):
  • Study Protocol (2020-11-22): https://cdn.clinicaltrials.gov/large-docs/56/NCT03160456/Prot_001.pdf